CLINICAL TRIAL: NCT01805167
Title: Electrophysiological Study of Interindividual Differences in Speech-understanding Among Cochlear Implant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-AOI-06; 2012-A01374-39 (Other: ANSM)
Record Dates: First submitted 2013-02-22; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-02

CONDITIONS: Hearing Loss
Keywords: Subject with cochlear implant
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- subjects with a cochlear implant (Other)
  Interventions: Other: Electrophysiological study of the interindividual variability of vocal performance

INTERVENTIONS:
Other: Electrophysiological study of the interindividual variability of vocal performance

SUMMARY:
Differences in speech-understanding and the quality of the subjective perception among cochlear implant patients (Digisonic SP) depends on numerous factors. The electrical field distribution (interaction between electrodes) could also explain the disparity of the performances? The objective of our study was to quantify the influence of the electrical field interactions between the channels of stimulation according to the vocal performances of the implanted subjects, for various subjective levels of electric stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject of French language
* Subject with a moderate bilateral sensorineural hearing loss, severe to profound
* Sensorineural hearing loss post-lingual (after onset of language acquisition)
* Subject paired with the implant Neurelec (Appendix 1) for more than 9 months
* Subject has received an appropriate setting under usual clinical follow-up
* Elderly 18 to 75 years
* Subject giving consent

Exclusion Criteria:

* Sensorineural hearing loss pre-lingual
* Deafness following a meningitis, or neurodegenerative diseases
* Illiteracy
* Pregnant women
* Subject blind
* Subject enjoying a measure of legal protection
* Subject incapable of giving consent
* Subject vulnerable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Quantify the interactions between electrical stimulation channels based vocal performance of implanted subjects, for different subjective levels of electrical stimulation. | At the inclusion - Day 0
  The vocal performance will be noted in percentage of voice recognition in the silence and in the noise.
  And the electric interaction between the channels of stimulations will be estimated by the measure of the refractory period of the circuits of the hearing system with the PEAEP after stimulations of electrodes of intermediate situation in the cochlée (electrodes 11, 12 and 13)

SECONDARY OUTCOMES:
Comparative study of PEAEP (Auditory Evoked Potentials Early electric) in vocal performance | At the inclusion - Day 0
  Collection of the PEAEP after stimulation of 4 different electrodes distributed on the totality of door-electrode: generally, electrodes 4, 7, 10 and 13 will be stimulated. The amplitudes and the latencies of the waves II, III and V will be analyzed and compared with the vocal performances.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guevara, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Guevara N, Hoen M, Truy E, Gallego S. A Cochlear Implant Performance Prognostic Test Based on Electrical Field Interactions Evaluated by eABR (Electrical Auditory Brainstem Responses). PLoS One. 2016 May 5;11(5):e0155008. doi: 10.1371/journal.pone.0155008. eCollection 2016. PMID 27149268